CLINICAL TRIAL: NCT02335008
Title: The Effect of Artificial Sweeteners (AFS) on Sweetness Sensitivity and Preference - Pilot Study
Brief Title: The Effect of Artificial Sweeteners (AFS) on Sweetness Sensitivity and Preference - Pilot
Acronym: AFS_pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Dana M. Small, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0405026766-1
Record Dates: First submitted 2014-10-24; First posted 2015-01-09 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Impairment of Oral Perception
MeSH Terms: interventions — trichlorosucrose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucralose (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with sucralose.
  Interventions: Dietary Supplement: Sucralose
- Sucrose (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with sucrose.
  Interventions: Dietary Supplement: Sucrose

INTERVENTIONS:
Dietary Supplement: Sucralose — 2 packets per 12 fl oz
  Arms: Sucralose
Dietary Supplement: Sucrose — equisweet to sucralose
  Arms: Sucrose

SUMMARY:
The goal of this study is to test the hypothesis that repeated consumption of artificial sweetener reduces sweet taste intensity.

DETAILED DESCRIPTION:
Significant controversy surrounds the possibility that consumption of artificial sweeteners (AFS) leads to weight gain. Some studies have found correlations between AFS use and weight gain and/or diabetes [1-4] while others have indicated that AFSs may aid in weight loss [5] or have no effects on body mass index (BMI) [6]. In rats, exposure to AFS leads to reduced chow intake following a sweet preload [7, 8], higher body weight [9, 10] and increased glucose responses and decreased GLP1 release following an oral glucose tolerance test [11] compared to exposure to caloric sweeteners. Given that the five FDA approved AFSs are found in thousands of foods [12] this marks a clear and significant gap in knowledge. Our preliminary data demonstrate a 3-fold decrease in sweet taste sensitivity following consumption of a beverage sweetened with two packets of Splenda for just 10 days. These data provide strong evidence that repeated exposure to sucralose reduces perception of sweet taste intensity, most likely by down-regulation of the sweet taste receptor. Therefore, it is imperative that we gain a greater understanding of the consequences of AFS use, since alterations in sweet taste perception that occur in response to AFS exposure may promote weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Fluent in English

Exclusion Criteria:

* History of oral nerve damage,
* presence of known taste or smell disorder,
* food allergies or sensitivities (for example nuts, lactose, artificial sweeteners),
* history of CNS disease,
* diabetes,
* history of DSM-IV major psychiatric disorder, including alcohol and substance abuse, chronic use of medication that may affect taste,
* conditions that may interfere with gustatory or olfactory perception (colds, seasonal allergies, recent smoking history),
* aberrant stimulus ratings,
* contra-indication for fMRI,
* uncomfortable swallowing in supine position.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Ratings of taste sensitivity | up to one week after intervention
  general labeled magnitude scale ratings of taste intensity

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, Principal Investigator — The John B Pierce Laboratory, Yale University
Locations (1):
- The John B Pierce Laboratory, New Haven, Connecticut, United States